CLINICAL TRIAL: NCT01483781
Title: A Double-Blind, Placebo-Controlled, Randomized, Parallel-Groups Study to Investigate the Effects of JNJ-28431754 (Canagliflozin) on Plasma Volume and Renal Function in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study of the Effects of Canagliflozin on Plasma Volume in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR100685; 28431754DIA1047 (Other: Janssen Research & Development, LLC); 2011-004117-17 (EudraCT Number)
Record Dates: First submitted 2011-11-30; First posted 2011-12-01 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Type 2; Plasma Volume
Keywords: Diabetes Mellitus, Type 2; Plasma Volume; Canagliflozin; Metformin; Hemoglobin A1c; Hypertension; Angiotensin-Converting Enzyme Inhibitors (ACEIs); Angiotensin Receptor Blockers (ARBs); Pharmacodynamics; Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Canagliflozin (Experimental)
  Interventions: Drug: Canagliflozin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin — Type = exact number, unit = mg, number = 300, form = capsule, route = oral use. One encapsulated tablet once daily for up to approximately 85 days (approximately 12 weeks)
  Arms: Canagliflozin
Drug: Placebo — Form = capsules, route = oral use. One capsule once daily for up to approximately 85 days (approximately 12 weeks)
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effects of canagliflozin on plasma volume and renal parameters in patients with Type 2 Diabetes Mellitus who are currently taking metformin and being treated for high blood pressure.

DETAILED DESCRIPTION:
This is a double-blind (neither the patient or study staff will know the identity of the treatment assigned) in patients with Type 2 Diabetes Mellitus (T2DM) who have inadequate glycemic (blood sugar) control on metformin monotherapy (metformin taken alone for control of T2DM) and who are currently being treated for hypertension (high blood pressure) with agents called angiotensin converting enzyme inhibitors (ACEIs) or angiotensin receptor blockers (ARBs). In the study, patients will be randomized (assigned by chance) to receive treatment with canagliflozin or a placebo (a treatment identical in appearance to canagliflozin but does not contain active drug) for 12 weeks. During the 12-week treatment period, patients will also take metformin at a dose of at least 1500 mg/day in addition to their prescribed ACEI or ARB for hypertension. Patients will participate in the study for up to approximately 22 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of T2DM with inadequate glycemic control (ie, HbA1c of >=7.0% and <=9.0% at Screening) on metformin monotherapy and be receiving therapy with an antihypertensive agent (an ACEI or ARB) for at least 4 weeks prior to Screening

Exclusion Criteria:

-History of diabetic ketoacidosis, type 1 diabetes mellitus (T1DM), pancreas or beta cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy; or a severe hypoglycemic episode within 6 months before screening

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in plasma volume (PV) | Baseline to Week 12 of the double-blind treatment period
  Baseline is defined as up to 3 days predose (Week -1)
Number of patients who experience at least 1 occurrence of a treatment-related adverse event | Day 1 to Day 85
  Treatment-related adverse events are adverse events with onset during the treatment phase.
Number of hypoglycemic events reported | Baseline up to Day 98
  Baseline is defined as up to 3 days predose (Week -1)
Change in electrocardiogram (ECG) parameters | Baseline up to Day 98
  Baseline is defined as up to 3 days predose (Week -1)
Change in blood pressure measurements | Baseline up to Day 98
  Baseline is defined as up to 3 days predose (Week -1)
Number of patients with physical examination findings reported as adverse events | Baseline up to Week 12
  Baseline is defined as up to 3 days predose (Week -1)
Change from baseline in pulse rate (beats/minute) | Baseline up to Day 98
  Baseline is defined as up to 3 days predose (Week -1)
Change in chemistry laboratory analytes | Baseline up to Day 98
  Baseline is defined as up to 3 days predose (Week -1)
Change from baseline in urinalysis laboratory analytes | Baseline up to Day 98
  Baseline is defined as up to 3 days predose (Week -1)
Change in hematology laboratory analytes | Baseline up to Day 98
  Baseline is defined as up to 3 days predose (Week -1)

SECONDARY OUTCOMES:
Change in PV | Baseline to Week 1 of the double-blind treatment period
  Baseline is defined as up to 3 days predose (Week -1)
Change in body weight | Baseline to approximately Week 1 and Week 12 of Double-Blind Treatment Phase
  Baseline is defined as up to 3 days predose (Week -1)
Change in 24-hour urine volume | Baseline to approximately Week 1 and Week 12 of Double-Blind Treatment Phase
  Baseline is defined as up to 3 days predose (Week -1)
Change in 24-hour fractional and total excretion of uric acid | Baseline to approximately Week 1 and Week 12 of Double-Blind Treatment Phase
  Baseline is defined as up to 3 days predose (Week -1)
Change in urine pH | Baseline to approximately Week 1 and Week 12 of Double-Blind Treatment Phase
  Baseline is defined as up to 3 days predose (Week -1)
Change in percent Hemoglobin A1c (HbA1c) | Baseline to Week 12
  Baseline is defined as up to 3 days predose (Week -1)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC L.L.C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: A Double-Blind, Placebo-Controlled, Randomized, Parallel-Groups Study to Investigate the Effects of JNJ-28431754 (Canagliflozin) on Plasma Volume and Renal Function in Subjects With Type 2 Diabetes Mellitus — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3346&filename=CR100685_CSR.pdf